CLINICAL TRIAL: NCT04504097
Title: Tushirikiane (Supporting Each Other): Development, Implementation and Evaluation of Novel HIV Self-Testing Delivery Approaches With Urban Displaced and Refugee Adolescents and Youth in Uganda
Brief Title: Tushirikiane HIV-self Testing Intervention With Urban Refugee Youth in Kampala, Uganda
Acronym: Tushirikiane
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Carmen Logie, MSW, PhD, Associate Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: CIHR389142
Record Dates: First submitted 2020-07-30; First posted 2020-08-07 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: HIV/AIDS; HIV Infections; Knowledge, Attitudes, Practice
Keywords: HIV self testing; Forcibly displaced youth; mhealth; HIV prevention; Uganda; informal settlements; linkage to confirmatory testing; routine HIV testing; HIV status knowledge; HIV care
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections; Behavior | interventions — American Recovery and Reinvestment Act

STUDY DESIGN:
Intervention Model Description: This cluster randomized controlled trial (cRCT) will evaluate the effectivness of HIVST delivery approaches on HIV testing uptake among refugee youth in Kampala. Clusters include 3 sites, informal settlements. Sites will be randomized in a 1:1:1 method to one of 3 study arms: Arm 1-HIVST, Arm 2- HIVST+ m-health, and Arm 3-standard of care (control). We propose a cRCT design of randomizing by slums to reduce the possibility of experimental contamination due to the shared social and physical environment in slums. Data collectors will administer tablet-based surveys (baseline, t1: 8 months, t2: 12 months). Arms 1 & 2 will receive HIVST kits at each time-point.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HIV self-testing + m-Health (Experimental): At the first visit participants will receive a HIVST kit and a detailed description of how to use the HIVST kits, pictorial and written guide for HIVST kits, condoms and lubricant, in addition to contact information for confirmatory testing and linkage to care at MARPI clinics. We will provide a 24-hour contact number to text, managed through WelTel system that will flag these messages in real-time. Participants will also receive a weekly bidirectional SMS hosted by WelTel to check how they are.
  Interventions: Behavioral: m-Health; Diagnostic Test: HIV self-testing
- HIV self-testing (Active Comparator): At the first visit participants will receive a HIVST kit and a detailed description of how to use the HIVST kits, pictorial and written guide for HIVST kits, condoms and lubricant, in addition to contact information for confirmatory testing and linkage to care at MARPI clinics
  Interventions: Diagnostic Test: HIV self-testing
- Standard of Care (No Intervention): Participants will receive information about HIV testing, care and support services at MARPI clinics and provide a pamphlet of information about HIV & HIV prevention strategies.

INTERVENTIONS:
Behavioral: m-Health — Participants receive a weekly bidirectional text message (SMS) asking how they are doing. They are requested to reply fine, or not fine, in which case they will be contacted with support by a peer navigator. If they do not reply to the message within the specified timeframe a peer navigator will follow up with them.
  Arms: HIV self-testing + m-Health
Diagnostic Test: HIV self-testing — Participants will receive HIVST kits so that they can perform their HIV testing.
  Arms: HIV self-testing; HIV self-testing + m-Health

SUMMARY:
HIV is the leading cause of death for adolescents and young people (AYP) in sub-Saharan Africa (SSA). Uganda hosts 1.3 million refugees/displaced persons, and more than 80,000 live in Kampala, most in slums, yet little is known of HIV testing and prevention needs with displaced/refugee AYP living in Kampala's slums. This study aims to develop, implement and evaluate an oral HIV-self testing (HIVST) intervention with displaced/refugee AYP aged 16- 24 in Kampala. HIVST is acceptable and properly used with AYP in other SSA regions, yet there are knowledge gaps regarding the best way to link HIVST to HIV care. This study aims to explore how m-health (healthcare delivered on mobile-phones), congruent with how AYP learn and socialize, can improve linkage to care with HIVST. This trial focuses on implementing a cluster randomized trial with displaced/refugee AYP aged 16-24 living in informal settlements in Kampala (Arm1: HIVST; Arm 2: HIVST + m-health; Arm 3: standard of care). The study will assess changes in HIV testing practices, HIV status knowledge, and linkage to HIV prevention and care between the 3 arms.

DETAILED DESCRIPTION:
The proposed study will take place in Kampala, Uganda, hosting over 80,000 refugees. This research will be conducted in 5 informal settlements ('slums') grouped into 3 clusters based on proximity (1: Kabalanga and Kasanga, 2: Katwe and Nsambya, 3: Rubaga) where most displaced/refugee persons in Kampala live.

The proposed intervention involves a cluster randomized controlled trial (cRCT) to evaluate the effectivness of HIVST delivery approaches on HIV testing uptake among refugee youth aged 16-24 in Kampala. Clusters include 3 sites, slums of: Kabalanga/kasanga, Katwe/Nsambya and Rubaga. Sites will be randomized in a 1:1:1 method to one of 3 study arms:

Arms 1 & 2: HIVST Interventions: At the first visit study participants are provided with a HIVST kit (Oraquick: approved and used in Uganda by the Ministry of Health) that is an oral swab test stick and tube solutions, and a written detailed step by step description of how to correctly use the HIVST kits, pictorial and written guide for HIVST kits, condoms and lubricant, information booklets on HIV and testing, referral cards with addresses and phone numbers to MARPI clinics for confirmatory testing. The cards will also have a peer navigator (PN)'s phone numbers for participants to text message (SMS) if they need additional information on how to use the kits, or support to go to confirmatory tests at the MARPI clinics. Instructions for the kits are in French, Swahili, Luganda and English and reflect the context of the urban displaced adolescent and young people. There is a 24-hour contact number for participants to text if/when they have questions. These texts will be managed through WelTel system that will flag these messages in real-time. The Research Coordinator and PN team will rotate being on-call to respond to these issues by text and will offer to phone, text, or WhatsApp support the participant and offer to make an appointment to see them and/or support them to attend MARPI or collaborating agency for further support. At follow-up visits PN will check in with participants about the HIVST kits, distribute another HIVST kit and condoms/lubricant, and screen for adverse events (e.g. negative HIVST related experiences).

Arm 2: HIVST + m-Health: Participants will receive weekly text messages via WelTel that check in with their wellbeing. Arm 2 PNs will discuss the weekly two-ways messages with participants, and request participants to respond to the message (detailed above) within 2 days.

Arm 3: Standard of Care: PNs will provide information about HIV testing, care and support services at MARPI clinics and provide a pamphlet of information about HIV & HIV prevention strategies (written in French, English, Luganda and Swahili).

Participant retention: Community collaborators will facilitate recruitment and retention; PNs will use multiple study reminder strategies (e.g. social media, texts) to maintain engagement, and we will utilize existing outreach and services by MARPI, YARID, Interaid Uganda, Tomorrow Vijana and community partners.

Research Team Training: This research involves collaborations with the Ministry of Health's Most At Risk Population Initiative (MARPI) clinics, YARID's women empowerment centre, Tomorrow Vijana's and Interaid Uganda's urban outreach programs in Kampala. MARPI clinic staff will provide technical assistance for HIVST and train PN and the research team in: a) using HIV rapid test kits (Alere Determine HIV-1/2); b) using OraQuick, a rapid oral HIVST used in Uganda; c) pre/post HIV test counseling; and d) linkages to confirmatory testing and HIV care.

m-Health training: This research involves a collaboration with WelTel's non-profit agency for the supportive SMS intervention (Arm 2). WelTel staff will conduct SMS training with: Research Coordinator, Logie, Okumu, and the research team, including the PN. The WelTel system will manage the SMS intervention on their structured mobile-phone platform (all SMS interactions are logged). Weekly 2-way supportive messages (how are you? In Swahili: Habari Yako?) will automatically be sent on the same weekday with WelTel software to Arm 2 participants. PN ask Arm 2 participants to respond within 48 hours if they are well (Mzuri sana) or have a problem (Nina shida), and will follow-up with non-responders. The Arm 2 PN and Research Coordinator will access the server every 24-48 hours to triage and respond to participants who express a problem or need.

Linkage to testing and care: Participants across all study arms will meet with PN at 3 time points (t0: baseline, t1: 8 months, t2: 12 months) to complete surveys. Each participant will have a study identification (ID) number printed on 'movie coupons'; they can bring these coupons to MARPI for HIV testing, confirmatory testing, linkage to HIV care, SRH services. The survey ID will be linked to resources accessed. Persons who test positive will be linked with the collaborator Uganda Network of Young People Living with HIV & AIDS (UNYPA)'s support groups and services.

ELIGIBILITY:
Inclusion Criteria:

* live in one of the 5 slum/informal settlement sites (Kabalanga, Kasanga, Katwe, Nsambya Rubaga)
* identify as a refugee/displaced person or have refugee parents
* aged 16-24
* report HIV negative status at baseline
* own or have access to a mobile phone for the study.

Exclusion criteria:

* report HIV-positive status at baseline
* do not identify as refugee or do not have refugee parents have no mobile phone do not live in the 5 selected slums

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 454 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
Changes in HIV testing Frequency | Time 1 (month 0), Time 2 (month 9), Time 3 (month 12)
  To assess changes in past 3 month HIV testing frequencies, participants are asked to self-report when their last HIV test was and where their last HIV test was (if they used the HIVST, clinic, or point-of-care testing).
Change in Knowledge of HIV status | Time 1 (month 0), Time 2 (month 9), Time 3 (month 12)
  To address social desirability bias challenges regarding self-reported HIV serostatus there are multiple steps employed. First, at Time 1 and Time 2 participants are asked their current HIV status.
  Second, participants are offered a completely voluntary rapid HIV test (Alere). Knowledge of HIV status will be assessed as correct for persons who agree to take the rapid test and correctly report their HIV status.
Changes in Linkage to confirmatory HIV testing | Time 2 (month 9), Time 3 (month 12)
  For arms 1 & 2 participants at Time 2 and Time 3 are asked if they used their HIVST kit; for those who respond affirmatively they will be asked the result, and those who report a positive result will be asked if and where they received confirmatory testing.
Changes in Linkage to HIV care | Time 2 (month 9), Time 3 (month 12)
  Participants who seroconvert during the study are asked the frequency of accessing HIV care services.
HIVST kit use | Time 3 (month 12)
  To understand the frequency of kit use by m-health arm, and to reduce social desirability bias regarding HIVST kit use, Arm 1 & 2 participants will be followed up one month after T3 to request to purchase unused kits back. Participants will not be informed of this as an option prior to this time.

SECONDARY OUTCOMES:
Changes in HIV stigma | Time 1 (month 0), Time 2 (month 9), Time 3 (month 12)
  HIV stigma outcomes will be assessed using Steward et al.'s 10 item perceived HIV stigma sbuscale. Higher scores indicate higher stigma.
Changes in Safer Sex Self-Efficacy. | Time 1 (month 0), Time 2 (month 9), Time 3 (month 12)
  Safer sex efficacy will be assessed using the Safer Sex Self-Efficacy Scale. Higher scores mean a better outcome. Range 5-20.
Changes in Consistent Condom Use Frequency. | Time 1 (month 0), Time 2 (month 9), Time 3 (month 12)
  Frequency of self-reported consistent condom use frequency (always vs. not always) will be assessed.
Changes in Sexual Relationship Power | Time 1 (month 0), Time 2 (month 9), Time 3 (month 12)
  Sexual relationship power will be assessed using the 15-item Relationship Control Sub-scale from the Sexual & Relationship Power Scale (SRPS). Scores range from 15-60. Higher scores mean a worse outcome.
Changes in adolescent sexual and reproductive health stigma. | Time 1 (month 0), Time 2 (month 9), Time 3 (month 12)
  Adolescent sexual and reproductive health (SRH) stigma will be assessed using the Adolescent SRH Stigma scale, sub-scale of sexual activity and pregnancy (7 items). Higher scores indicate higher stigma.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Logie, PhD, Principal Investigator — University of Toronto, Canada
Locations (1):
- Factor-Inwentash Faculty of Social Work, University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
The final dataset will consist of self-reported demographic and social-ecological data from interviews with the participants and laboratory data from HIV confirmatory tests for HIV positive individuals. Even though the final dataset will be de-identified before release for sharing, it may be possible to deductively disclose subjects using a combination of common characteristics. Therefore, to access our data, users need to meet our data-sharing agreement that provides for: (1) ability to secure ethics approval from both the user's institution and the University of Toronto research ethics board (2) a commitment to using the data solely for research purposes and not to identify any individual participant; (3) a dedication to securing the data using appropriate computer technology such as encryption; and (4) a commitment to destroying or returning the data after analyses are completed.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 1 year after final data collection time point.
Access Criteria: (1) ability to secure ethics approval from both the user's institution and the University of Toronto research ethics board (2) a commitment to using the data solely for research purposes and not to identify any individual participant; (3) a dedication to securing the data using appropriate computer technology such as encryption; and (4) a commitment to destroying or returning the data after analyses are completed.

REFERENCES:
- [Derived] Logie CH, Okumu M, Berry I, Hakiza R, Baral SD, Musoke DK, Nakitende A, Mwima S, Kyambadde P, Loutet M, Batte S, Lester R, Neema S, Newby K, Mbuagbaw L. Findings from the Tushirikiane mobile health (mHealth) HIV self-testing pragmatic trial with refugee adolescents and youth living in informal settlements in Kampala, Uganda. J Int AIDS Soc. 2023 Oct;26(10):e26185. doi: 10.1002/jia2.26185. PMID 37850816
- [Derived] Logie C, Okumu M, Hakiza R, Kibuuka Musoke D, Berry I, Mwima S, Kyambadde P, Kiera UM, Loutet M, Neema S, Newby K, McNamee C, Baral SD, Lester R, Musinguzi J, Mbuagbaw L. Mobile Health-Supported HIV Self-Testing Strategy Among Urban Refugee and Displaced Youth in Kampala, Uganda: Protocol for a Cluster Randomized Trial (Tushirikiane, Supporting Each Other). JMIR Res Protoc. 2021 Feb 2;10(2):e26192. doi: 10.2196/26192. PMID 33528378